CLINICAL TRIAL: NCT02672202
Title: Shifting Pain Modulation From Pro-to Anti-nociceptive: Individualized Prevention of Post Operative Pain
Brief Title: Shifting Pain Modulation From Pro-to Anti-nociceptive
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment rate was slow so we could not complete the study.
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 614-15-RMB Hernia_CTIL
Record Dates: First submitted 2016-01-12; First posted 2016-02-03 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Post-operative Chronic Pain
Keywords: Chronic Pain; Pain Modulation Profile; CPM; acute post operative pain
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain | interventions — Duloxetine Hydrochloride; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Duloxetine (Active Comparator): Treatment
  Interventions: Drug: Duloxetine; Drug: Placebo
- Pregabalin (Active Comparator): Treatment
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — * 60 mg/d - twice before surgery and once a day for post operative days 3-7
  * 30 mg/d - once a day for post operative days 1-2
  Arms: Duloxetine
Drug: Pregabalin — * 75 mg/d - twice a day for post operative days 1-2
  * 150 mg/d - twice a day for post operative days 3-7 300 mg/d - twice before surgery
  Arms: Pregabalin
Drug: Placebo — * non-active - twice before surgery
  * non-active - twice a day for post operative days 1-7
  Arms: Duloxetine; Placebo

SUMMARY:
To create a data base that will facilitate the enrichment of the insights regarding post-operative pain development, and to identify those individuals with the potential to develop this kind of pain. The identification will be based on the individualized pain modulation profile, composed of a battery of tests as detailed below.

DETAILED DESCRIPTION:
Background

Pro-nociceptive pain modulation profile (PMP) is characterized by either:

(i) decreased inhibition of pain, i.e.inhibitory pro-nociceptive PMP, (ii) increased facilitation, i.e. facilitatory pro-nociceptive PMP, or (iii) both, i.e. dual pro-nociceptive PMP.

The counterpart of pro-nociceptive, i.e., anti-nociceptive PMP, has not yet been explored. The investigators expect individuals harboring this profile to be at lower risk for pain acquisition, and experience less intense pain. Pain modulation is commonly altered in pain patients toward a pro-nociceptive pain modulation profile (PMP), expressed, in the lab, by increased facilitation and/or decreased inhibition of experimental pain, and clinically by high pain phenotype.

The proposed study seeks to explore the yet to be characterized mirror image of pro-nociception, i.e., the situation where individuals exhibit reduced pain facilitation and more efficient pain inhibition. This domain of 'anti-nociceptive' PMP is a potential platform for improving pain therapy and prevention. Extrapolating from the clinical picture of pro-nociception, it is likely that 'antinociceptive' individuals will express a lower pain phenotype, with less frequent and less intense pain experiences, lower risk of acquiring pain after surgery or trauma, and, possibly, better response to analgesics. The investigators would like to explore whether it is possible to shift pain modulation towards anti-nociception, in order to obtain the possible benefits of this modulation profile in pain-prone situations.

The clinical model the investigators propose for addressing the hypotheses is preemptive drug treatment for reduction of postoperative pain. Our specific choice of surgery is inguinal herniorraphy. In addition to acute post-operative pain, this operation carries a relatively high rate of chronic post-operative pain (ranging from 10 to 54% of patients, with most reports indicating towards the lower end of this range).

Our specific aims are to explore, in the setup of post operative pain after inguinal herniorraphy, the shift of PMP from pro- towards anti-nociceptive based on each of the following testing domains:

(i) Psychophysical and neurophysiological data describing facilitatory and inhibitory modulation capacity of the patient.

(ii) Psychological data describing patient's behavior such as catastrophizing, anxiety and depression, pain sensitivity and life orientation.

(iii) Blood tests to evaluate Micro RNA which regulate downstream transcription or shutting down gene expression, in order to evaluate their role as predictor for evolving chronic pain, and (v) individual case data related to age, gender, education, socioeconomic parameters and personal medical history.

Subjects

* Study A: One hundred and forty healthy subjects (range 20-79; 20 subjects per age decade, 10 M, and 10 F) will participate in the first phase of the study aimed to collect normative data from healthy population.
* Study B: Two hundred and twenty patients (range 18-75) scheduled for inguinal herniorraphy will be enrolled.

Study design Study I - Normative data collection for the inhibitory and excitatory pain modulation responses, a study on healthy subjects

The study will include one session. In this session, after signing informed consent, subjects will:

(i) fill out state of health questionnaire, (ii) record 5 minutes of resting state EEG, and (iii) undergo a short familiarization with the various stimulation modalities.

Thereafter, and along the session subjects will fill the pain related personality questionnaires (anxiety and depression, catastrophizing, pain sensitivity, life orientation test and ten item personality measure) followed by psychophysical assessments, which will include assessment of conditioned pain modulation (CPM) and temporal pain summation (TS) as described later on. A sample of 20 ml of blood will be drawn from all subjects at the end of the session.

Study II - Herniorraphy surgery patients This study is a randomized, placebo-controlled, double-blind, three parallel arms non-crossover longitudinal study in four groups of patients identified by their PMPs. The study will consist of two assessment sessions: the first between 1 to 2 weeks before surgery and the second 3 month after surgery. The sessions will be conducted by experienced experimenter, and will include the same psychophysical and psychological assessments as in Study I; after signing informed consent, patients will undergo a short familiarization with the various stimulation modalities and then undergo the various stimuli.

At the end of this session patients will be assigned into one of four groups:

(i) dual pro-nociceptive, (ii) inhibitory pro-nociceptive, (iii) facilitatory pro-nociceptive, and (iv) anti-nociceptive.

45 patients will be assigned into each group, by order of their recruitment. Third of the patients in each group will be randomized to Duloxetine (DUL), third to Pregabalin (PGB) and the other third to Placebo (PLA). Each group will receive two treatment doses of the drug before surgery, i.e. one in the evening before and one at the morning of the surgery. Patients will then undergo surgery, to be performed by one team of surgeons, under a standardized protocol of general anesthesia. After surgery patients will be treated by a standardized analgesic protocol until discharge, normally the morning after surgery. Acute pain intensity and analgesics consumption during the first 24 hours will be recorded. On post-operative day (POD) 1 patients will fill a "patient outcome questionnaire" that will include information about their perceived post-operative pain intensity and the extent of pain interference with activities and effects on mood and anxiety. A periodic phone call for chronic postoperative pain will be pursued at 1, 2, 4 weeks and 6 months after surgery. An experimenter blinded to the psycho-physical group assignment, will follow the pain state after surgery.

Two samples of 20 ml of blood will be drawn from all patients; first blood withdrawal will be done before surgery, and the second at a clinic visit between 3 and 6 month after surgery.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists (ASA) I - III patients planned for elective herniorraphy.

Exclusion Criteria:

* Report of pain at hernia site for more than 30 on 0-100 Numeric Pain Scale (NPS) (ranging from 0, denoting ''no pain'', to 100, denoting ''the worst pain imaginable''), for most of the days during past one month.
* Regular use of analgesia for any purpose, including serotonin-norepinephrine re-uptake inhibitors (SNRIs) and gabapentins during the previous month.
* Use of monoamine oxidase inhibitors (MAOIs) within the last 14 days.
* Narrow-angle glaucoma.
* Known pregnancy or lactation.
* Chronic pain disorders.
* Inability to perform psycho-physical testing, as in the case of cognitive or psychiatric disorders. Participants will sign a consent form before recruitment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-02; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change in pain scores as measured by numerical pain scale (NPS) | 6 months
  Change in post-operative pain - acute post operative pain transform into chronic pain. A periodic phone call will be pursued at 1, 2, 4 weeks and 6 months after surgery
Therapeutic response to the analgesic drugs | 48 hours
  The level of the pain relief. Acute post-operative pain measured by analgesic consumption during hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: David Yarnitsky, Principal Investigator — Head of Neurology department at Rambam